CLINICAL TRIAL: NCT05781191
Title: Analysis of the Determinants of Refusal and Adherence to Coadministration of Influenza Vaccination With the Booster of COVID-19 Vaccine on Health Care Workers of the Fondazione Policlinico Universitario "A. Gemelli" IRCCS
Brief Title: Analysis of the Determinants of Adherence to Coadministration of Flu Vaccination With the Booster of COVID-19 Vaccine
Acronym: CoVFlu
Status: Completed | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Laurenti Patrizia, Chief of the Complex Operative Unit of Hospital Hygiene, University Polyclinic Foundation "A. Gemelli" IRCCS, Rome, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 5169
Record Dates: First submitted 2023-03-10; First posted 2023-03-23 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Influenza; COVID-19
MeSH Terms: conditions — Influenza, Human; COVID-19 | interventions — BNT162 Vaccine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Employees
  Interventions: Biological: COMIRNATY

INTERVENTIONS:
Biological: COMIRNATY — Booster (3rd) dose of COMIRNATY Seasonal dose of influenza vaccination based on patient's individual risk factors
  Other Names: FLUAD TETRA; FLUCELVAX TETRA; FLUARIX TETRA

SUMMARY:
This study investigates healthcare workers' attitudes towards co-administering COVID-19 and seasonal influenza vaccines, a method supported globally for its efficiency and potential to lessen healthcare burdens. It explores various factors affecting workers' willingness to accept or decline this approach, ranging from demographic to logistical aspects, and examines the link between vaccine hesitancy and co-administration acceptance, aiming to identify and address hesitancy towards both vaccines

DETAILED DESCRIPTION:
Analysis of the determinants of refusal and adherence to the coadministration of influenza vaccination with the booster dose of anti-SARS-CoV-2 vaccine conducted on healthcare personnel of the University Polyclinic Foundation "A. Gemelli" IRCCS New evidence now suggests that co-administration of COVID-19 vaccines with inactivated vaccines is acceptable in terms of immunogenicity and reactogenicity. In particular, a recent randomized placebo-controlled phase IV study, established that both ChAdOx1 and BNT162b2 COVID-19 vaccines could be safely co-administered with seasonal influenza (SIV) vaccines adjuvanted with MF59 or derived from cell culture, without any clinically significant increase in adverse events or immunologic inference.

Although limited data are available, Interim Guidelines issued by WHO suggest that such co-administration is acceptable. The U.S. Centers for Disease Control and Prevention (CDC) supports that COVID-19 vaccines can be co-administered with other vaccines, including SIV. Similarly, in October 2021 (i.e., just before the start of the 2021/2022 flu vaccination campaign), the Italian Ministry of Health gave the go-ahead for co-administration of the vaccine.

Vaccination programs against COVID-19 and seasonal influenza are currently being implemented in parallel in many countries. The administration of both vaccines during the same session would have several advantages. At the individual level, it would reduce the number of necessary health visits and provide timely protection against both diseases; these individual benefits may encourage greater uptake of the two vaccines. Also from the perspective of health system organization and management, co-administration could facilitate the implementation of both vaccine programs and reduce the overall burden on health services.

The primary objective of the study is to measure the modifiable and non-modifiable, subjective and objective, demographic, economic, social, cultural, occupational, logistical and personal determinants of refusal or adherence to co-administration of seasonal influenza vaccination with the booster dose of anti-SARS-CoV vaccine-Evaluate the association between refusal of co-administration and vaccine hesitancy, both general and specific for influenza and/or SARS-cov-2;

1. Identify subgroups most at risk of refusing co-administration;
2. Identify the most appropriate interventions and/or incentives to overcome the main determinants of refusal to co-administer;
3. Identify the most appropriate interventions and/or incentives to overcome the main determinants of co-administration refusal.

ELIGIBILITY:
Inclusion Criteria:

* All healthcare workers and non-employees of FPG and all Physicians in Specialty Training attached to UCSC will be enrolled during the period when the possibility of coadministration of the two vaccines (Sars-CoV-2 and influenza) was available at the Foundation at the Covid-19 Vaccine Center set up at Presidio Columbus and/or at specially designated facilities, i.e., between November 13, 2021 and December 31, 2021.

Exclusion Criteria:

* All individuals who have received vaccinations, influenza and/or anti-SARS-CoV-2 with booster dose, outside the window in which coadministration was available at FPG will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will have an expected duration of 6 months from the date of Ethics Committee approval. The data analyzed will refer to the period: November 13, 2021-December 31, 2021.
Sampling Method: Non-Probability Sample
Enrollment: 8231 (Actual)
Dates: Start 2021-11-13 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Determinants of refusal of co-administration | 31-12-2021
  Modifiable and nonmodifiable subjective and objective demographic, economic, social, cultural, occupational, logistical, and personal determinants of refusal or adherence to coadministration of seasonal influenza vaccination with the booster dose of anti-SARS-CoV-2 vaccine

SECONDARY OUTCOMES:
Association with vaccine hesitancy | 31-12-2021
  Association between refusal of coadministration and vaccine hesitancy, both general and specific for influenza and/or SARS-CoV-2;
Sub-groups at risk | 31-12-2021
  Identify the subgroups most at risk of refusing co-administration;
Most appropriate interventions | 31-12-2021
  Identify the most appropriate interventions and/or incentives to overcome the main determinants of refusal to co-administer;

CONTACTS AND LOCATIONS:
Overall Officials: Patrizia Laurenti, MD, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli IRCCS - Rome
Locations (1):
- Fondazione Policlinico Gemelli, Roma, RM, Italy

IPD SHARING:
Plan to Share IPD: No